CLINICAL TRIAL: NCT02954094
Title: A Longitudinal Observational Study of the Natural History and Management of Patients With Hepatocellular Carcinoma
Brief Title: A Longitudinal Observational Study of the Natural History and Management of Patients With HCC
Status: Active, not recruiting | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-HCC
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Patients enrolled in TARGET-HCC may be invited to participate in the Biorepository Specimen Bank (BSB). Blood samples and tissue samples for biomarker and DNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study. These samples will be shipped to a central repository for storage to use in future studies. Samples stored at the biorepository will be identified only with the participant's unique study ID number and the date that the sample was obtained. This link between the participant's study ID number and their name will be available only at the site where the samples were obtained.
Oversight: Data Monitoring Committee: No

SUMMARY:
TARGET-HCC is a longitudinal, observational study of patients being managed for HCC in usual clinical practice. TARGET-HCC will create a research registry of participants with HCC within academic and community real-world practices in order to assess the safety and effectiveness of the entire spectrum of current and future therapies across diverse populations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age ≥18 years
2. Patients with a histological/cytological or radiological diagnosis of HCC (mixed HCC cholangiocarcinoma may be included; patients who are candidates for surgical and non-surgical treatment, as well as those being followed without specific HCC therapy may be included)

Exclusion Criteria:

1. Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients being managed for HCC
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Establish a longitudinal observational cohort to understand the natural history and management of HCC, including the safety and outcomes of HCC treatment interventions utilized in usual clinical practice | Up to 15 years

SECONDARY OUTCOMES:
Evaluate the impact of HCC treatment interventions and concomitant medications on comorbid conditions and liver function | Up to 15 years
Evaluate patient-reported outcomes measures during the natural course of HCC and management with HRQoL questionnaires | Up to 15 years
Establish a Biorepository Specimen Bank (BSB) | Up to 15 years

CONTACTS AND LOCATIONS:
Locations (71):
- United States (52):
  - Banner University Medical Center, Phoenix, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - University of Southern California/Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California-Davis, Sacramento, California
  - University of California, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - Gastro Florida, Clearwater, Florida
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - University of Florida Health Gastroenterology, Jacksonville, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Division of Gastroenterology and Hepatology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - Mercy Medical Center, GI Research, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research (STAR) LLC, Jackson, Mississippi
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Northwell Health - Center for Liver Diseases, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Center for Liver Disease and Transplant at CMC, Charlotte, North Carolina
  - Providence Health & Services Cancer Clinical Trials, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center - GI Research Office, Nashville, Tennessee
  - Clinical Research Institute@ Methodist Dallas Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott & White All Saints, Fort Worth, Texas
  - Research Specialists of Texas, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - University of Wisconsin, Madison, Wisconsin
- France (2):
  - CHU de Nice - Hôpital L'Archet 2, Nice
  - Hôpitaux Universitaires Paris Centre, Paris
- Germany (8):
  - Universitätsklinikum Aachen, Aachen
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz
- Italy (4):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - A.O.U.P. di Palermo, Palermo
  - Humanitas Mirasole IRCCS, Rozzano
  - IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo
- Spain (5):
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabrera R, Singal AG, Colombo M, Kelley RK, Lee H, Mospan AR, Meyer T, Newell P, Parikh ND, Sangro B, Reddy KR, Watkins S, Zink RC, Di Bisceglie AM. A Real-World Observational Cohort of Patients with Hepatocellular Carcinoma: Design and Rationale for TARGET-HCC. Hepatol Commun. 2020 Dec 21;5(3):538-547. doi: 10.1002/hep4.1652. eCollection 2021 Mar. PMID 33681685